CLINICAL TRIAL: NCT03508999
Title: Effectiveness of Metronidazole Gel and Mobile Telephone Short- Message Service Reminders on Gingivitis in Orthodontic Patients: A Randomized Controlled Trial
Brief Title: Effectiveness of Metronidazole Gel and Mobile SMS Reminders on Gingivitis in Orthodontic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Hafiz Taha Mahmood, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gingivitis_Orthodontics
Record Dates: First submitted 2018-03-29; First posted 2018-04-26 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metronidazole Gel (Experimental): Group A subjects will be given standard oral hygiene instructions on the visit with a standard 0.8 % metronidazole gel instructed to apply topically on the marginal gingiva for the next 4 weeks, twice a day for 30 minutes, after morning and evening tooth brushing.
  Interventions: Drug: Metronidazole gel
- SMS Text Reminder (Other): Subjects will be provided biweekly reminder via SMS in the form of text message reinforcing oral hygiene. Additionally, patients will be given standard oral hygiene instructions on the visit with a placebo gel topically instructed to apply on the marginal gingiva for the next 4 weeks, twice a day for 30 minutes, after morning and evening tooth brushing.
  Interventions: Other: SMS text reminder
- Placebo (Placebo Comparator): Group C will be subjects will be given standard oral hygiene instructions on the visit with a placebo gel topically instructed to apply on the marginal gingiva for the next 4 weeks, twice a day for 30 minutes, after morning and evening tooth brushing.
  Interventions: Other: Placebo gel

INTERVENTIONS:
Drug: Metronidazole gel — The application of metronidazole gel is effective in the management of gingivitis in patients undergoing orthodontic therapy. Additionally, the constant reminder therapy at weekly interval would also lead to improvement in the oral hygiene.16 According to pertinent literature survey, none of the study has been conducted to compare the effectiveness of SMS reminders and use of anaerobic gel to reduce gingival inflammation.
  Other Names: Anaerobic gel
  Arms: Metronidazole Gel
Other: SMS text reminder — Subjects will be provided biweekly reminder via 'SMS text reminder' in the form of text message reinforcing oral hygiene. Additionally, patients will be given standard oral hygiene instructions on the visit with a placebo gel topically instructed to apply on the marginal gingiva for the next 4 weeks, twice a day for 30 minutes, after morning and evening tooth brushing.
  Other Names: Reminder
  Arms: SMS Text Reminder
Other: Placebo gel — Group C will be subjects will be given standard oral hygiene instructions on the visit with a placebo gel topically instructed to apply on the marginal gingiva for the next 4 weeks, twice a day for 30 minutes, after morning and evening tooth brushing.
  Arms: Placebo

SUMMARY:
A rapid deterioration in oral hygiene occur after bonding of orthodontic appliances. Zachrisson and Zachrisson have reported that even after maintaining excellent oral hygiene, patients usually experience mild to moderate gingivitis within 1-2 months after orthodontic appliance placement. Slutzkey and Levin have reported a prevalence of 72 % gingivitis in orthodontic patients.

The difficulty in maintenance of oral hygiene and inefficient removal of supragingival plaque due to the appliances lead to development of gingivitis and hyperplasia. Tooth brush access to the buccal surface of the teeth becomes problematic and predisposes plaque buildup around the brackets.

Investigators are now focusing on the development of localized drug delivery systems that can allow maximum concentration on the target site, thus minimizing the potential systemic effects. Metronidazole has been used by several researchers due to its selective antimicrobial activity against the obligate anaerobes. The topical administration in gel form has several advantages. Miani et al concluded that the use of metronidazole gel significantly reduces the total bacterial count in the gingival crevicular fluid.

In medicine and dentistry, active mobile telephone short-message service (SMS) reminders have been used to improve patient compliance and positive behavior changes. A study conducted by Epprighta et al have reported the effectiveness of SMS reminder in orthodontic patients. They have reported significantly lower bleeding, gingival and plaque indices scores in SMS reminder group as compared to control.

Rationale:

The application of metronidazole gel is effective in management of gingivitis in patients undergoing orthodontic therapy. Additionally, the constant reminder therapy at weekly interval would also lead to improvement in the oral hygiene. According to pertinent literature survey, none of the study has been conducted to compare the effectiveness of SMS reminders and use of anaerobic gel to reduce gingival inflammation.

Null Hypothesis:

Application of 0.8% metronidazole gel and mobile telephone short-message service oral hygiene reminders is equally effective in reducing the gingival inflammation in orthodontic patients with gingivitis as compared to control group.

Objective:

The objectives of the study will be to assess the use of topical gel or mobile telephone short-message service oral hygiene reminders can reduce gingivitis in orthodontic patients as compared to control group.

DETAILED DESCRIPTION:
Gingivitis: It is defined as the inflammation of the gingiva in the absence of clinical attachment loss.

Six standard sites on incisors, canines and premolars have been used in this study as study sites as described by Gettinger et al. The investigators will not include banded first molars because the banding itself will lead to a compromise in periodontal conditions. The study sites will be six proximal-buccal line angles on the following teeth: right maxillary second premolar, mesiobuccal line angle; right maxillary canine, distobuccal line angle; left maxillary central incisor, distolabial line angle; right mandibular central incisor, distolabial line angle; left mandibular canine, distobuccal line angle; and left mandibular second premolar, mesiobuccal line angle. If a study tooth was missing, the corresponding tooth on the contralateral side was examined. All study sites will be evaluated at baseline (To) and 4 weeks later at (T1).

Bleeding Index (BI): BI will be scored as described by Saxton and van der Ouderaa upon probing the gingival sulci of six standard sites mentioned above.

0. Absence of bleeding after 30 seconds

1. Bleeding observed after 30 seconds
2. Immediate bleeding

Gingival index:

0. No inflammation.

1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.

Orthodontic Plaque Index (PI):

According to Orthodontic Plaque Index, the investigators will assess the six standard sites and the condition of adjacent marginal gingiva by staining the teeth with plaque disclosing solution (erythrosine).

0. No plaque deposits on the tooth surfaces surrounding the bracket base

1. Plaque deposits on one tooth surface at the bracket base
2. Plaque deposits on two tooth surface at the bracket base
3. Plaque deposits on three tooth surface at the bracket base
4. Plaque deposits on four tooth surface at the bracket base and/or gingival inflammation indicators (plaque deposits near the gingiva do not necessarily have to be present) Study Setting: Dental clinic, Aga Khan University Hospital, Karachi Duration Of Study: Four months after approval of synopsis by Ethical Review Committee of AKU

Sample Size:

Sample size is calculated in OpenEpi (version 3.01) sample size calculator. Martin et al reported that the mean gingival index at 4-6 weeks interval in gel group was 1.56 + 0.14; while in the control group, it was 1.68 + 0.12.

Keeping the above difference at the level of significance (α) at 5% and power of study (1-β) at 95%, the investigators need at least 19 observations for each arm. The sample size is inflated by 10% to get 21 subjects per arm for any loss to follow up or noncompliance to metronidazole/placebo gel.

Since, the investigators have three experimental groups, so the investigators need a total of 63 subjects.

Sampling Technique: Random Permuted block sampling 6 and 8

Ethical considerations:

The study will be started after obtaining approval from ethical review committee. Only those participants will be recruited who will sign the consent form. The study will be conducted according to the World Medical Association's Declaration of Helsinki and the principles of GCP (Good Clinical Practice). Any subsequent protocol amendments will be submitted to ERC and regulatory authorities for approval. The trial will be conducted in compliance with regulations, particularly specifying pharmaco-vigilance reporting and a copy of final study report will be submitted to ERC.

Possible Risks or Benefits:

There may be no risk involved in this study as the study is based on treatment options which is routinely used in dental clinics to treat gingivitis. The metallic taste in the metronidazole gel might lead to nausea.

Benefits include the evaluation of the best modality to manage gingivitis in orthodontic patients. Additionally, there would not be any direct benefit to the participants but significant results from the study would lead to improvement in the standard protocol for future patients.

Adverse Events:

There is no adverse event reported in the literature related to topical gel to be used in the study. The trial related events would be covered by the department of surgery. The product related adverse events would be managed, reported and recorded to ERC within a specified period of time while the serious adverse events will be reported immediately to ERC.

Right Of Refusal To Participate And Withdrawal:

Participants will be given choice to either participate or refuse to participate in the study All participants non-compliant with gel therapy will be excluded from the study

Incentive:

After T1 all patients will be given free of cost scaling and polishing treatment. If the indices are still high, and clinical examination shows higher score of gingivitis, additional systemic antibiotics will be prescribed.

Patient confidentiality, access and storage:

The information provided by the participant will remain confidential. Nobody except investigators will have access to it. Participants' name and identity will not be disclosed at any time. However, the data may be seen by ethical review committee, DSMB or any local regulatory body. As per GCP and other guidelines, data will be retained for 15 years.

Randomization, blinding and treatment allocation:

Subjects will be assigned to one of the three study groups using a computer generated randomization list. The randomization will be performed by clinical trials unit (CTU) using a random permuted block sampling of 6 and 8. The study investigators will be blinded and only CTU pharmacist will be unblinded in this study.

The recruitment of the patients will be performed by one investigator who will explain the objective and three arms of the study and participant could be in any arm that is selected by computer. All the measurements at the baseline (To) and follow ups (T1) will be recorded by the second investigator on separate To and T1 sheets. Patient and the investigator who is taking the measurement will be blinded about the intervention groups. The reminder SMS messages will be sent by another clinician who will not be the part of the study.

Investigational product management:

The metronidazole gel 0.8% contains metronidazole tablets and carboxy methyl cellulose 2% as a base solution. The placebo gel contains similar ingredients except metronidazole tablet. The metronidazole and placebo gel will be prepared by Pharmacy Department, Aga Khan University Hospital. The participants will be instructed to apply 1.5 gm approximately metronidazole/placebo gel (Aga Khan University Hospital) twice daily for four weeks. The participants will be given tubes of metronidazole/placebo gel each stored at room temperature. The packing, labelling, storage and dispatch of the gel will be performed by clinical trials unit.

Data collection procedure:

Ethical approval will be taken from the institutional ethical review committee before commencement of the study. All those patients who fulfilled the inclusion criteria will receive detailed information regarding the study and only those patients will be included who signed an informed consent.

Training of the examiner:

Participating investigator will be trained and calibrated on the development of the trial, case selection, measurement techniques, sample collection, data compilation sheets and their precise role in the study. For assessment of intra-examiner reliability, measurements will be repeated by same investigator for 5 subjects at 1 week interval.

Data analysis:

Data will be analyzed using SPSS version 20.0. Descriptive statistics for all the base line clinical parameters such as bleeding index, orthodontic plaque index and gingival index scores will be calculated. It will be an intention to treat analysis. Gingival index, bleeding index and orthodontic plaque index will be compared across group A, B and C. The level of significance will be kept at < 0.05.

Finance:

Department of Surgery

Publication policy/plan:

The data will be used for the publication nationally and internationally and could be presented in either local or international forum.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthodontic treatment with fixed appliance since 6 months
* Patients with all bonded teeth mesial to the first molars and not adjacent to a banded tooth
* Systematically healthy patient with no co-morbid such as rheumatic fever, blood dyscrasias, congenital heart disease or diabetes mellitus
* Subjects with gingivitis as assessed by bleeding index (score =2), orthodontic plaque index (score ≥ 2) and gingival index (score ≥ 2) as assessed by Williams Probe
* All patients who sign the inform consent will be included in the study

Exclusion Criteria:

* Subjects with clinical attachment loss of greater than 2 mm on two sites
* Pregnant or lactating females
* Subjects with removal or fixed dental prosthesis, teeth with banding used for attachment
* History of surgical or nonsurgical periodontal therapy in the last 6 months
* Use of antibiotic or anti-inflammatory in the last 30 days confirmed by patient's history
* Habit of smoking or use of smokeless tobacco
* Allergic to Metronidazole according to patient history

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Improvement of Bleeding Index | Improvement in Bleeding Index Scores at 4 Weeks
  Improvement in Bleeding Index Scores In Orthodontic Patients, Change from Baseline in Index at 4 weeks. All the measurements at the baseline (To) and follow ups (T1) will be recorded by the investigator on separate To and T1 sheets. Six standard sites on incisors, canines and premolars have been used in this study as study sites. The study sites will be six proximal-buccal line angles on the following teeth: right maxillary second premolar, mesiobuccal line angle; right maxillary canine, distobuccal line angle; left maxillary central incisor, distolabial line angle; right mandibular central incisor, distolabial line angle; left mandibular canine, distobuccal line angle; and left mandibular second premolar, mesiobuccal line angle. If a study tooth was missing, the corresponding tooth on the contralateral side will be examined.
  0. Absence of bleeding after 30 seconds
  1. Bleeding observed after 30 seconds
  2. Immediate bleeding
Improvement in Gingival index | Improvement in Gingival Index Scores at 4 Weeks
  Improvement in Gingival Index Scores In Orthodontic Patients, Change from Baseline in Index at 4 weeks. All the measurements at the baseline (To) and follow ups (T1) will be recorded by the investigator on separate To and T1 sheets. Six standard sites on incisors, canines and premolars have been used in this study as study sites (same as above).
  0. No inflammation.
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding
Improvement of Orthodontic Plaque Index | Improvement in Orthodontic Plaque Index Scores at 4 Weeks
  Improvement in Orthodontic Plaque Index Scores In Orthodontic Patients, Change from Baseline in Index at 4 weeks. All the measurements at the baseline (To) and follow ups (T1) will be recorded by the investigator on separate To and T1 sheets. Six standard sites on incisors, canines and premolars have been used in this study as study sites (same as above) and the condition of adjacent marginal gingiva by staining the teeth with plaque disclosing solution will be assessed.
  0. No plaque deposits on the tooth surfaces surrounding the bracket base
  1. Plaque deposits on one tooth surface at the bracket base
  2. Plaque deposits on two tooth surface at the bracket base
  3. Plaque deposits on three tooth surface at the bracket base
  4. Plaque deposits on four tooth surface at the bracket base and/or gingival inflammation indicators (plaque deposits near the gingiva do not necessarily have to be present)

CONTACTS AND LOCATIONS:
Overall Officials: Mubassar Fida, BDS, FCPS, Principal Investigator — Consultant
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Jewair TS, Suri S, Tompson BD. Predictors of adolescent compliance with oral hygiene instructions during two-arch multibracket fixed orthodontic treatment. Angle Orthod. 2011 May;81(3):525-31. doi: 10.2319/092010-547.1. Epub 2011 Feb 9. PMID 21306222
- [Background] Timmerman MF, van der Weijden GA. Risk factors for periodontitis. Int J Dent Hyg. 2006 Feb;4(1):2-7. doi: 10.1111/j.1601-5037.2006.00168.x. PMID 16451433
- [Background] Zachrisson S, Zachrisson BU. Gingival condition associated with orthodontic treatment. Angle Orthod. 1972 Jan;42(1):26-34. doi: 10.1043/0003-3219(1972)0422.0.CO;2. No abstract available. PMID 4500561
- [Background] Slutzkey S, Levin L. Gingival recession in young adults: occurrence, severity, and relationship to past orthodontic treatment and oral piercing. Am J Orthod Dentofacial Orthop. 2008 Nov;134(5):652-6. doi: 10.1016/j.ajodo.2007.02.054. PMID 18984397
- [Background] O'Reilly MM, Featherstone JD. Demineralization and remineralization around orthodontic appliances: an in vivo study. Am J Orthod Dentofacial Orthop. 1987 Jul;92(1):33-40. doi: 10.1016/0889-5406(87)90293-9. PMID 3300270
- [Background] Lundstrom F, Krasse B. Caries incidence in orthodontic patients with high levels of Streptococcus mutans. Eur J Orthod. 1987 May;9(2):117-21. doi: 10.1093/ejo/9.2.117. No abstract available. PMID 3472889
- [Background] Alexander SA. The effect of fixed and functional appliances on enamel decalcifications in early Class II treatment. Am J Orthod Dentofacial Orthop. 1993 Jan;103(1):45-7. doi: 10.1016/0889-5406(93)70103-U. PMID 8422030
- [Background] Ainamo J. Control of plaque by chemical agents. J Clin Periodontol. 1977 Dec;4(5):23-35. doi: 10.1111/j.1600-051x.1977.tb00049.x. No abstract available. PMID 275277
- [Background] Hanes PJ, Purvis JP. Local anti-infective therapy: pharmacological agents. A systematic review. Ann Periodontol. 2003 Dec;8(1):79-98. doi: 10.1902/annals.2003.8.1.79. PMID 14971250
- [Background] Slots J, Ting M. Systemic antibiotics in the treatment of periodontal disease. Periodontol 2000. 2002;28:106-76. doi: 10.1034/j.1600-0757.2002.280106.x. No abstract available. PMID 12013339
- [Background] Loesche WJ. Antimicrobials in dentistry: with knowledge comes responsibility. J Dent Res. 1996 Jul;75(7):1432-3. doi: 10.1177/00220345960750070101. No abstract available. PMID 8876593
- [Background] Pavia M, Nobile CG, Bianco A, Angelillo IF. Meta-analysis of local metronidazole in the treatment of chronic periodontitis. J Periodontol. 2004 Jun;75(6):830-8. doi: 10.1902/jop.2004.75.6.830. PMID 15295949
- [Background] Miani PK, do Nascimento C, Sato S, Filho AV, da Fonseca MJ, Pedrazzi V. In vivo evaluation of a metronidazole-containing gel for the adjuvant treatment of chronic periodontitis: preliminary results. Eur J Clin Microbiol Infect Dis. 2012 Jul;31(7):1611-8. doi: 10.1007/s10096-011-1484-7. Epub 2011 Dec 6. PMID 22138847
- [Background] Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med. 2009 Feb;36(2):165-73. doi: 10.1016/j.amepre.2008.09.040. PMID 19135907
- [Background] Eppright M, Shroff B, Best AM, Barcoma E, Lindauer SJ. Influence of active reminders on oral hygiene compliance in orthodontic patients. Angle Orthod. 2014 Mar;84(2):208-13. doi: 10.2319/062813-481.1. Epub 2013 Sep 12. PMID 24028316
- [Background] Gettinger G, Patters MR, Testa MA, Loe H, Anerud A, Boysen H, Robertson PB. The use of six selected teeth in population measures of periodontal status. J Periodontol. 1983 Mar;54(3):155-9. doi: 10.1902/jop.1983.54.3.155. PMID 6573472
- [Background] Saxton CA, van der Ouderaa FJ. The effect of a dentifrice containing zinc citrate and Triclosan on developing gingivitis. J Periodontal Res. 1989 Jan;24(1):75-80. doi: 10.1111/j.1600-0765.1989.tb00860.x. PMID 2524573
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Beberhold K, Sachse-Kulp A, Schwestka-Polly R, Hornecker E, Ziebolz D. The Orthodontic Plaque Index: an oral hygiene index for patients with multibracket appliances. Orthodontics (Chic.). 2012;13(1):94-9. PMID 22567620
- [Background] Martin BJ, Campbell PM, Rees TD, Buschang PH. A randomized controlled trial evaluating antioxidant-essential oil gel as a treatment for gingivitis in orthodontic patients. Angle Orthod. 2016 May;86(3):407-12. doi: 10.2319/041515-251.1. Epub 2015 Aug 17. PMID 26280662